CLINICAL TRIAL: NCT06554639
Title: A Phase 1, Open-Label, Fixed-Sequence Study to Evaluate the Effects of Multiple Doses of Diltiazem on the Single-Dose Pharmacokinetics of MK-5684 in Healthy Adult Male Participants
Brief Title: A Drug-Drug Interaction Study of Diltiazem and MK-5684 in Healthy Adult Male Participants (MK-5684-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5684-011; MK-5684-011 (Other: MSD)
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; fludrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-5684 Period 1 (Experimental): On Day 1 a single dose of MK-5684 will be administered under fasting conditions and a single dose of HRT (prednisone and fludrocortisone) will be administered under fed conditions approximately 4.5 hours after MK-5684 dosing.
  Interventions: Drug: MK-5684; Drug: Prednisone; Drug: Fludrocortisone acetate
- MK-5684 Period 2 (Experimental): There will be a washout of at least 5 days between MK-5684 dosing in Period 1 and the first diltiazem dosing in Period 2. In Period 2, diltiazem will be administered once daily (QD) for 6 consecutive days with a single dose of MK-5684 coadministered on Day 2 under fasting conditions. HRT (prednisone and fludrocortisone) will be administered under fed conditions QD on Days 2 through 5, approximately 4.5 hours after MK-5684 and/or diltiazem dosing.
  Interventions: Drug: MK-5684; Drug: Prednisone; Drug: Fludrocortisone acetate; Drug: Diltiazem hydrocholoride

INTERVENTIONS:
Drug: MK-5684 — Administered via oral tablet per dosing regimen.
Drug: Prednisone — Administered at a dose of 2.5 mg or 5 mg dependent on HRT dosing regimen via oral tablets.
Drug: Fludrocortisone acetate — Administered at a dose of 0.05 mg per HRT dosing regimen via oral tablets.
Drug: Diltiazem hydrocholoride — Administered at a dose of 240 mg per dosing regimen via oral capsule (extended-release).
  Arms: MK-5684 Period 2

SUMMARY:
Researchers have designed a study medicine called MK-5684 as a new way to treat prostate cancer.

The purpose of this study is to learn what happens to MK-5684 in a person's body over time (a pharmacokinetic or PK study). Researchers will compare what happens to MK-5684 in the body when it is given with and without another medicine called diltiazem.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m^2
* Able to swallow multiple tablets

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History or presence of any of the following:

  * Adrenal insufficiency
  * Hepatic or renal impairment
  * Clinically significant hypotension, cardiac arrhythmia, cardiac conduction abnormalities, or recurrent unexplained syncopal events
  * Second- or third-degree Atrioventricular (AV) heart block (except in participants with a functional artificial pacemaker)
  * Clinically significant sick sinus syndrome
  * Presence of any systemic fungal infection
  * Chronic infection
  * Glaucoma
  * Hypothyroidism
  * Stomach ulcer
  * Ocular herpes simplex
* Has a first-degree relative with multiple unexplained syncopal events, unexplained cardiac arrest, or sudden cardiac death, or has a known family history of an inherited arrhythmia syndrome (including Brugada syndrome)
* History of cancer (malignancy)
* Unable to refrain from or anticipants the use of: Unable to refrain from or anticipates the use of: Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from 0 to infinity after single dosing (AUC0-inf) of MK-5684 in plasma | Predose, and at designated timepoints up to 120 hours post-dose
  AUC0-inf of MK-5684 in plasma will be determined.
Area under the concentration versus time curve from 0 to last quantifiable sample (AUC0-last) of MK-5684 in plasma | Predose, and at designated timepoints up to 120 hours post-dose
  AUC0-last of MK-5684 in plasma will be determined.
Area under the concentration versus time curve from 0 to Hour 24 (AUC0-24) of MK-5684 in plasma | Predose, and at designated timepoints up to 24 hours post-dose
  AUC0-24 of MK-5684 in plasma will be determined.
Maximum concentration (Cmax) of MK-5684 in plasma | Predose, and at designated timepoints up to 120 hours post-dose
  Cmax of MK-5684 in plasma will be determined.
Time to Maximum concentration (Tmax) of MK-5684 in plasma | Predose, and at designated timepoints up to 120 hours post-dose
  Tmax of MK-5684 in plasma will be determined.
Apparent terminal half-life (t1/2) of MK-5684 in plasma | Predose, and at designated timepoints up to 120 hours post-dose
  t1/2 of MK-5684 in plasma will be determined.
Apparent Clearance (CL/F) of MK-5684 in plasma | Predose, and at designated timepoints up to 120 hours post-dose
  CL/F of MK-5684 in plasma will be determined.
Apparent volume of distribution during terminal phase (Vz/F) of MK-5684 in plasma | Predose, and at designated timepoints up to 120 hours post-dose
  Vz/F of MK-5684 in plasma will be determined.

SECONDARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to approximately 39 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to approximately 39 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/